CLINICAL TRIAL: NCT02618486
Title: The Effects of Obesity on Non Surgical Periodontal Therapy
Acronym: EONSPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101269-1
Record Dates: First submitted 2015-11-03; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Obese; Periodontal Disease
MeSH Terms: conditions — Obesity; Periodontal Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese with CP (Experimental): Procedure/Surgery Non surgical periodontal therapy Received OHE, scaling and root planing. OHE includes brushing and flossing techniques, chlorhexidine rinse thrice a day
  Interventions: Procedure: Non surgical periodontal therapy
- Non obese with CP (Active Comparator): Procedure/Surgery Non surgical periodontal therapy Received OHE, scaling and root planing. OHE includes brushing and flossing techniques, chlorhexidine rinse thrice a day
  Interventions: Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — NSPT includes oral hygiene education, scaling root planing and mouth wash
  Other Names: NSPT

SUMMARY:
The investigators' earlier study reported a high prevalence of chronic periodontitis among obese Malaysian adult population. Non-surgical periodontal therapy (NSPT) has been shown to effectively reduce microbial load and contributes to reduction in periodontal parameters and inflammatory burden up to 6 months post-therapy. This study will cast light on the effects of obesity on chronic periodontitis (CP) patients following NSPT. The objectives of the study were to quantify and to compare the periodontal pathogens, serum and salivary interleukins in obese and non obese with CP following NSPT.

DETAILED DESCRIPTION:
Obesity is a health concern, associated with complex diseases such as diabetes, hypertension as well as chronic periodontitis. The prevalence is estimated as 24% worldwide, 3% for South East Asia, and 27.2% for Malaysia. Prevalence of CP is increasing, with 10-15% reported in various adult populations and estimated 5-20% categorised as severe CP. In Malaysia, the prevalence of severe CP is estimated as 18%.

The first paper on the relationship between obesity and periodontal disease reported that obese-hypertensive rats are more likely to have periodontal tissue deterioration than normal rats. Subsequent study reported an induction of expression of Tumour Necrosis Factor (TNF) -a gene in obese mice and thus proposed TNF-α represents a key mediator of obesity-linked insulin resistance. This was strongly supported by an extension study on human adipose tissue. A model was proposed linking inflammation to obesity, diabetes, and periodontal infection in 2005. Subsequent studies found association between obesity and increased risk for CP in the United States, Japanese and Jordanian adult populations.

Adipose tissue produces a number of adipokines linked to inflammation, including adiponectin, interleukin (IL)-1β, IL-6, TNF-α, Monocyte Chemoattractant Protein (MCP)-1 and Macrophages Migrant Inhibitory Factor (MIF). Increased in circulating levels of pro-inflammatory cytokines such as TNF-α and IL-6 are strongly correlated with obesity, insulin resistance, hyperglycemia and diabetes mellitus. These cytokines also stimulate the synthesis of C-reactive protein (CRP) and fibrinogen by liver, as CRP is known for its role in inflammation, atherosclerosis and insulin resistance. In addition, these cytokines are also secreted from adipose tissues are involved in the pathophysiology of both obesity and periodontitis. Obese individuals have higher levels of circulating TNF-α and IL-6 when compared to normal weight individuals. This may increase the risk of destructive periodontal diseases development. Interestingly, studies on the immune response to periodontal pathogens showed that TNF-α enhanced the immune response to these pathogens.

Periodontal health is accomplished through non-surgical periodontal therapy (NSPT), which includes oral hygiene education (OHE) and scaling and root planing (SRP). NSPT has been reported to effectively reduce microbial load and contributes to reduction in periodontal parameters and inflammatory burden up to 6 months post-therapy. In a general population, NSPT has been shown to induce a shift from a pre-dominant gram-negative to a gram-positive subgingival microbiota. The total bacteria count and positives sites of Porphyromonas gingivalis (P gingivalis) and Tannerella forsythia (T forsythia) were significant decreased in treated group compared to control groups. In addition, SRP has markedly reduced these periodontal pathogens: Porphyromonas gingivalis, Tannerella forsythia as well as Prevotella intermedia 24 months post NSPT.

Molecular mechanisms between inflammatory cytokines and CP are unclear and warrant further studies to determine whether pro-inflammatory cytokines is the pathogenic factor linking obesity to periodontal infections. To date, there are not many studies that examine the changes in periodontal pathogen, salivary and serum interleukins levels in obese patients with CP following NSPT. Further prospective studies are needed to address this issue and to determine stronger evidence on the association between obesity, periodontal diseases and potential mediating factors following NSPT.

ELIGIBILITY:
Inclusion Criteria:

* Those who are obese
* Those whose age are 30 years and above
* Those who have at least 12 teeth present

Exclusion Criteria:

* Those who have received periodontal treatment within the last 4 months
* Those who have been on antibiotics within the past 4 months
* Those who require prophylactic antibiotic coverage, on systemic or topical steroidal anti-inflammatory drugs for the past 4 months,
* Those who are pregnant or intend to be pregnant
* Those lactating mothers, mentally handicapped

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in clinical attachment level (CAL) (mean in mm, as a measure of periodontal parameter) in obese and non obese, with chronic periodontitis following NSPT | 12 weeks

SECONDARY OUTCOMES:
Changes in microbial profile (mean count of Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia and Actinobacillus actinomycetemcomitans quality and quantity) in obese and non obese, with chronic periodontitis before and after NSPT | 12 weeks
Changes in serum interleukins levels (mean value in ng/mL, of TNF-α, IL-1, IL-6 and resistin) in obese and non obese, with chronic periodontitis before and after NSPT | 12 weeks
Changes in salivary interleukins levels (mean value in ng/mL, of TNF-α, IL-1, IL-6 and resistin) in obese and non obese, with chronic periodontitis before and after NSPT | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nor_Adinar Baharuddin, DClinDent, Principal Investigator — Faculty of Dentistry University of Malaya Kuala Lumpur

REFERENCES:
- [Background] Khan S, Saub R, Vaithilingam RD, Safii SH, Vethakkan SR, Baharuddin NA. Prevalence of chronic periodontitis in an obese population: a preliminary study. BMC Oral Health. 2015 Sep 29;15:114. doi: 10.1186/s12903-015-0098-3. PMID 26419358
- [Background] Albandar JM, Tinoco EM. Global epidemiology of periodontal diseases in children and young persons. Periodontol 2000. 2002;29:153-76. doi: 10.1034/j.1600-0757.2002.290108.x. No abstract available. PMID 12102707
- [Background] Albandar JM, Brunelle JA, Kingman A. Destructive periodontal disease in adults 30 years of age and older in the United States, 1988-1994. J Periodontol. 1999 Jan;70(1):13-29. doi: 10.1902/jop.1999.70.1.13. PMID 10052767
- [Background] Hugoson A, Norderyd O, Slotte C, Thorstensson H. Distribution of periodontal disease in a Swedish adult population 1973, 1983 and 1993. J Clin Periodontol. 1998 Jul;25(7):542-8. doi: 10.1111/j.1600-051x.1998.tb02485.x. PMID 9696253
- [Background] Brown LJ, Loe H. Prevalence, extent, severity and progression of periodontal disease. Periodontol 2000. 1993 Jun;2:57-71. doi: 10.1111/j.1600-0757.1993.tb00220.x. No abstract available. PMID 9673181
- [Background] Petersen PE, Bourgeois D, Ogawa H, Estupinan-Day S, Ndiaye C. The global burden of oral diseases and risks to oral health. Bull World Health Organ. 2005 Sep;83(9):661-9. Epub 2005 Sep 30. PMID 16211157
- [Background] Brennan DS, Spencer AJ, Roberts-Thomson KF. Quality of life and disability weights associated with periodontal disease. J Dent Res. 2007 Aug;86(8):713-7. doi: 10.1177/154405910708600805. PMID 17652197
- [Background] Petersen PE. The World Oral Health Report 2003: continuous improvement of oral health in the 21st century--the approach of the WHO Global Oral Health Programme. Community Dent Oral Epidemiol. 2003 Dec;31 Suppl 1:3-23. doi: 10.1046/j..2003.com122.x. PMID 15015736
- [Background] Mohamud WN, Musa KI, Khir AS, Ismail AA, Ismail IS, Kadir KA, Kamaruddin NA, Yaacob NA, Mustafa N, Ali O, Isa SH, Bebakar WM. Prevalence of overweight and obesity among adult Malaysians: an update. Asia Pac J Clin Nutr. 2011;20(1):35-41. PMID 21393108
- [Background] Kurukulasuriya LR, Stas S, Lastra G, Manrique C, Sowers JR. Hypertension in obesity. Med Clin North Am. 2011 Sep;95(5):903-17. doi: 10.1016/j.mcna.2011.06.004. PMID 21855699
- [Background] Park SH, Park JH, Song PS, Kim DK, Kim KH, Seol SH, Kim HK, Jang HJ, Lee JG, Park HY, Park J, Shin KJ, Kim Di, Moon YS. Sarcopenic obesity as an independent risk factor of hypertension. J Am Soc Hypertens. 2013 Nov-Dec;7(6):420-5. doi: 10.1016/j.jash.2013.06.002. Epub 2013 Jul 30. PMID 23910010
- [Background] Marotta T, Russo BF, Ferrara LA. Triglyceride-to-HDL-cholesterol ratio and metabolic syndrome as contributors to cardiovascular risk in overweight patients. Obesity (Silver Spring). 2010 Aug;18(8):1608-13. doi: 10.1038/oby.2009.446. Epub 2009 Dec 17. PMID 20019684
- [Background] Matsushita Y, Nakagawa T, Yamamoto S, Kato T, Ouchi T, Kikuchi N, Takahashi Y, Yokoyama T, Mizoue T, Noda M. Adiponectin and visceral fat associate with cardiovascular risk factors. Obesity (Silver Spring). 2014 Jan;22(1):287-91. doi: 10.1002/oby.20425. Epub 2013 Jun 11. PMID 23519992
- [Background] Rasmussen F, Hancox RJ. Mechanisms of obesity in asthma. Curr Opin Allergy Clin Immunol. 2014 Feb;14(1):35-43. doi: 10.1097/ACI.0000000000000024. PMID 24300417
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Perlstein MI, Bissada NF. Influence of obesity and hypertension on the severity of periodontitis in rats. Oral Surg Oral Med Oral Pathol. 1977 May;43(5):707-19. doi: 10.1016/0030-4220(77)90055-x. PMID 266151
- [Background] Al-Zahrani MS, Bissada NF, Borawskit EA. Obesity and periodontal disease in young, middle-aged, and older adults. J Periodontol. 2003 May;74(5):610-5. doi: 10.1902/jop.2003.74.5.610. PMID 12816292
- [Background] Khader YS, Bawadi HA, Haroun TF, Alomari M, Tayyem RF. The association between periodontal disease and obesity among adults in Jordan. J Clin Periodontol. 2009 Jan;36(1):18-24. doi: 10.1111/j.1600-051X.2008.01345.x. Epub 2008 Nov 19. PMID 19046327
- [Background] Trayhurn P, Wood IS. Adipokines: inflammation and the pleiotropic role of white adipose tissue. Br J Nutr. 2004 Sep;92(3):347-55. doi: 10.1079/bjn20041213. PMID 15469638
- [Background] Khosravi R, Ka K, Huang T, Khalili S, Nguyen BH, Nicolau B, Tran SD. Tumor necrosis factor- alpha and interleukin-6: potential interorgan inflammatory mediators contributing to destructive periodontal disease in obesity or metabolic syndrome. Mediators Inflamm. 2013;2013:728987. doi: 10.1155/2013/728987. Epub 2013 Aug 28. PMID 24068858
- [Background] Fentoglu O, Koroglu BK, Hicyilmaz H, Sert T, Ozdem M, Sutcu R, Tamer MN, Orhan H, Ay ZY, Ozturk Tonguc M, Kirzioglu FY. Pro-inflammatory cytokine levels in association between periodontal disease and hyperlipidaemia. J Clin Periodontol. 2011 Jan;38(1):8-16. doi: 10.1111/j.1600-051X.2010.01644.x. Epub 2010 Nov 10. PMID 21062339
- [Background] Noh MK, Jung M, Kim SH, Lee SR, Park KH, Kim DH, Kim HH, Park YG. Assessment of IL-6, IL-8 and TNF-alpha levels in the gingival tissue of patients with periodontitis. Exp Ther Med. 2013 Sep;6(3):847-851. doi: 10.3892/etm.2013.1222. Epub 2013 Jul 15. PMID 24137277
- [Background] Saxlin T, Ylostalo P, Suominen-Taipale L, Mannisto S, Knuuttila M. Association between periodontal infection and obesity: results of the Health 2000 Survey. J Clin Periodontol. 2011 Mar;38(3):236-42. doi: 10.1111/j.1600-051X.2010.01677.x. Epub 2010 Dec 27. PMID 21198765
- [Background] D'Aiuto F, Parkar M, Andreou G, Suvan J, Brett PM, Ready D, Tonetti MS. Periodontitis and systemic inflammation: control of the local infection is associated with a reduction in serum inflammatory markers. J Dent Res. 2004 Feb;83(2):156-60. doi: 10.1177/154405910408300214. PMID 14742655
- [Background] Ryan ME. Nonsurgical approaches for the treatment of periodontal diseases. Dent Clin North Am. 2005 Jul;49(3):611-36, vii. doi: 10.1016/j.cden.2005.03.010. PMID 15978244
- [Derived] Md Tahir K, Ab Malek AH, Vaithilingam RD, Saub R, Safii SH, Rahman MT, Abdul Razak F, Alabsi AM, Baharuddin NA. Impact of non-surgical periodontal therapy on serum Resistin and periodontal pathogen in periodontitis patients with obesity. BMC Oral Health. 2020 Feb 14;20(1):52. doi: 10.1186/s12903-020-1039-3. PMID 32059714